CLINICAL TRIAL: NCT05339126
Title: RNS System Feasibility Study of Thalamocortical Brain-Responsive Neurostimulation for the Treatment of Lennox-Gastaut Syndrome
Brief Title: RNS System LGS Feasibility Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroPace (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NP10015; UH3NS109557 (NIH)
Record Dates: First submitted 2022-03-29; First posted 2022-04-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy; Lennox Gastaut Syndrome; Lennox-Gastaut Syndrome, Intractable; Seizures; Seizures, Generalized
Keywords: Medically refractory; Responsive neurostimulation; RNS System; Thalamocortical stimulation
MeSH Terms: conditions — Epilepsy; Lennox Gastaut Syndrome; Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Condition A (Active Comparator): high-frequency short bursts (HFSB: 100 Hz, 160 µs pulse width, 200 msec burst)
  Interventions: Device: RNS System
- Condition B (Active Comparator): low-frequency long bursts (LFLB: 5 Hz, 160 µs pulse width, 5 sec burst)
  Interventions: Device: RNS System

INTERVENTIONS:
Device: RNS System — The RNS System provides closed loop responsive brain stimulation. The Neurostimulator monitors the electrical activity of the brain to detect abnormal activity that could lead to a seizure. If abnormal activity is detected, the neurostimulator delivers electrical stimulation to the brain through the leads to help prevent the seizure before it occurs.

SUMMARY:
To generate preliminary safety and effectiveness data for brain-responsive neurostimulation of thalamocortical networks as an adjunctive therapy in reducing the frequency of generalized seizures in individuals 12 years of age or older with Lennox Gastaut Syndrome (LGS) who are refractory to antiseizure medications.

The intent is to determine the feasibility and the optimal design of a subsequent pivotal study in order to expand the indication for use for the RNS System as a treatment for patients with medically intractable LGS.

DETAILED DESCRIPTION:
This study is a prospective two-stage single-blind feasibility cross-over study designed to provide early safety and preliminary evidence of effectiveness for combined bilateral brain-responsive neurostimulation of thalamocortical networks for the treatment of generalized seizures in patients with LGS. Twenty participants will be treated with the RNS System across six Comprehensive Epilepsy Centers in the U.S. Enrollment will be staged in two cohorts of 10. Once all 10 participants of the first cohort complete Treatment Block 1 and the interim analysis criteria are met, the next cohort of 10 participants will be enrolled. The research study comprises six study periods:

1. Baseline Period
2. Implant (surgery)
3. Post-Op Period
4. Blinded Evaluation Period (which is made up of 3 treatment blocks, one of which is a sham stimulation)
5. Open Label Period
6. Long Term Follow-Up Period

Two neurostimulators will be placed: one in the parieto-temporal skull on the left, and the second in the homologous region on the right. Depth leads will target the bilateral CM. Cortical strip or depth leads will target the prefrontal cortex. Each neurostimulator will be connected to two ipsilateral leads: one in the prefrontal cortex and one in the CM. A total of two neurostimulators and four leads will be implanted. During the Blinded Evaluation Period, the participant will move through 3 different treatment blocks (Treatment Block1, Treatment Block 2, and Treatment Block 3) in a random order. Two of the blocks will have active stimulation treatment and one of the blocks will have no (sham) stimulation treatment. The participant and caregiver will be blinded to the treatment condition.

* Condition A - active treatment of high frequency short burst stimulation
* Condition B - active treatment of low frequency long burst stimulation
* Sham - no stimulation treatment

After completing the Blinded Evaluation Period the participant will transition to the 1-year Open Label Period and have study appointments every 3 months. After completing the 1-year Open Label Period the participant will transition to the Long Term Follow-up Period. The Long-Term Follow-up Period may last up to 2 years with appointments every 3 months until the participant complete this research or this research study ends.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 15 years of age or older for first cohort; 12 years of age or older for second cohort. Note that age requirements for eligibility differ by cohort, as follows: the age limit for Cohort 1 is 15 years of age and above and the age limit for Cohort 2 may decrease to 12 years, pending a DSMB letter of recommendation, based on review of interim data analysis and concurrence with NINDS.
* Participant has medically intractable epilepsy defined as failure to achieve acceptable seizure control without unacceptable medication related side effects despite trials of 2 or more antiseizure medications.
* Participant had an average of ≥ 5 drop seizures per month in the 2 months preceding enrollment. A drop seizure is defined as an epileptic seizure (atonic, tonic, tonic-clonic, or myoclonic) involving the entire body, trunk, or head that leads or could lead to a fall, injury, or slumping in a chair.
* Participant's seizures are non-localized.
* Participant's scalp recorded EEG has features of LGS, such as multifocal spike, slow spike and wave discharges, and paroxysmal fast activity.
* Participant must (a) have a stable antiseizure medication (ASM) regimen for the 2 months preceding enrollment and (b) be willing to remain on the stable regimen, as medically able, through the Blinded Evaluation Period; rescue medication for acute seizure clusters are permitted. A stable ASM regimen is defined as no introduction or discontinuation of an ASM, and no change in an ASM dose of more than 25%.
* Participant is not on a therapeutic diet for epilepsy, or if participant is on a therapeutic diet for epilepsy must (a) have a stable diet for the 2 months preceding enrollment and (b) be willing to remain on the stable diet, as medically able, through the Blinded Evaluation Period.
* Participant does not have a vagus nerve stimulator (VNS), or if participant does have a VNS must (a) have had the VNS off for the 2 months preceding enrollment and (b) be willing to remain with the VNS off through the Blinded Evaluation Period.
* Participant is a male, or is a female of childbearing potential who is surgically sterile, 2 years postmenopausal, or practices a reliable method of contraception (hormonal, barrier method or abstention).
* Participant is willing to give informed consent (or assent, if a minor); if the participant assents or is not able to give informed consent, parent/legal guardian is willing to give informed consent.
* Participant is able to maintain a seizure log alone or with the assistance of a competent individual.
* Participant is able to attend study appointments in accordance with the study schedule.

Exclusion Criteria:

* Participant is participating in a therapeutic investigational drug or device study (including other RNS System studies).
* Participant is currently implanted with an electronic medical device that delivers electrical energy to the brain.
* Participant is currently implanted with an RNS Neurostimulator or NeuroPace Leads.
* Participant requires procedures that are contraindicated based on current RNS System labeling.
* Participant is pregnant.
* Participant has a diagnosed unstable psychiatric disorder or any attempt or expressed intent of suicide over the preceding 6 months.
* In the opinion of the investigator, the participant has a clinically significant or unstable medical condition [including alcohol, opioid, recreational cannabis (not for therapeutic purposes) or other drug use disorder] or a progressive central nervous system disease.
* Participant is taking any anticoagulants.
* In the opinion of the investigator, participant is an unsuitable candidate for this procedure.
* Participant has been diagnosed with psychogenic or non-epileptic seizures in the preceding year.
* Participant has experienced unprovoked status epilepticus in the preceding year.
* Participant has had therapeutic surgery to treat epilepsy in the preceding 3 months. Participants who have had epilepsy surgery more than 3 months prior to enrollment are eligible.

Note: For contraindications, refer to current physician labeling (manuals) for the RNS System available at the NeuroPace website (www.neuropace.com).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Annual device-related serious adverse event (SADE) rate | 12 months post-implant
  The lower limit of the 95% confidence interval of the annual SADE rate at months 12 and 24 post-implant is less than 33.6% and 22.0%, respectively (twice the SADE rate of 16.8% and 11.0%, respectively, at the same time points in the RNS System pivotal study)
Safety: Annual device-related serious adverse event (SADE) rate | 24 months post-implant
  The lower limit of the 95% confidence interval of the annual SADE rate at months 12 and 24 post-implant is less than 33.6% and 22.0%, respectively (twice the SADE rate of 16.8% and 11.0%, respectively, at the same time points in the RNS System pivotal study)
Effectiveness: Blinded evaluation period (BEP) responder rate | 12 months post-implant
  The responder rate during one or both of the stimulation conditions (A or B) is ≥ 30%.
  The responder rate is the proportion of participants that are responders. A responder in this study is defined as a participant who has a ≥ 35% reduction in the frequency of drop seizures compared to that participant's pre-implant baseline.

SECONDARY OUTCOMES:
Safety: Post-op SAE rate | 4 weeks post-implant
  The lower limit of the 95% confidence interval of the SAE rate following the implant procedure (through 4 weeks post-op) is less than 24% (twice the SAE rate of 12% at the same time point in the RNS System pivotal study).

OTHER OUTCOMES:
Rate of SAEs of particular relevance | Every 12 months post-implant
  The annual event rate of SAEs of particular relevance (device-related or not) will be calculated over time of study participation. SAEs of particular relevance include those related to: death, erosion, infection, suicidality, depression, hemorrhage, seizure-related injury, and tolerability of stimulation
Affective status | Implant through 4 years post-implant
  Affective status (by summary scores from the Beck Depression Inventory, either the BDI-II or BYI-II, depending on age at time of the initial clinic appointment) will be described for the pre-implant baseline, as well as at the transition to Treatment Block 1, Treatment Block 2, Treatment Block 3, and Open Label; and for every 6 months thereafter that the participant is in the study.
Cognitive function | Implant through 2 years post-implant
  Neuropsychological functioning as assessed by neuropsychological testing with validated, standardized inventories to assess domains that include attention (Flanker Inhibitory Control and Attention Test). The inventory is taken from the NIH Toolbox Cognition Battery and will be described by presenting summary scores for the pre-implant baseline, as well as for the end of the Blinded Evaluation Period and for the end of the Open Label Period.
Cognitive function | Implant through 2 years post-implant
  Neuropsychological functioning as assessed by neuropsychological testing with validated, standardized inventories to assess three domains that include memory (Picture Sequence Memory Test). The inventory is taken from the NIH Toolbox Cognition Battery and will be described by presenting summary scores for the pre-implant baseline, as well as for the end of the Blinded Evaluation Period and for the end of the Open Label Period.
Cognitive function | Implant through 2 years post-implant
  Neuropsychological functioning as assessed by neuropsychological testing with validated, standardized inventories to assess three domains that include vocabulary (Picture Vocabulary Test). The inventory is taken from the NIH Toolbox Cognition Battery and will be described by presenting summary scores for the pre-implant baseline, as well as for the end of the Blinded Evaluation Period and for the end of the Open Label Period.
Median percent change in seizure counts | Implant through 4 years post-implant
  Median percentage change in counts of:
  * Drop seizures, and
  * Tonic-clonic seizures during both stimulation conditions (A and B), and every year thereafter while participating in the study, compared to that participant's pre-implant baseline
Days with seizures | Implant through 4 years post-implant
  Days with:
  * Any type of seizure
  * Drop seizures
  * Non-drop seizures during pre-implant baseline, during both stimulation conditions (A and B), and every year thereafter while participating in the study.
  A non-drop seizure is defined as an absence seizure, a myoclonic seizure, or an atonic or tonic seizure not leading to a fall.
Participant quality of life as measured by the QOLIE-AD-48 | Implant through 4 years post-implant
  Quality of life for the pre-implant baseline, as well as at the transitions to Treatment Block 1, Treatment Block 2, Treatment Block 3, and Open Label; and for every 6 months thereafter that the participant is in the study according to the QOLIE-AD-48 (validated for ages 12-17 years, depending on age at time of assessment).
Participant quality of life as measured by the QOLIE-31-P | Implant through 4 years post-implant
  Quality of life for the pre-implant baseline, as well as at the transitions to Treatment Block 1, Treatment Block 2, Treatment Block 3, and Open Label; and for every 6 months thereafter that the participant is in the study, according to the QOLIE-31-P (validated for ages 18 and older, depending on age at time of assessment).
Caregiver burden | Implant through 4 years post-implant
  Caregiver burden for the pre-implant baseline, as well as at the transitions to Treatment Block 1, Treatment Block 2, Treatment Block 3, and Open Label; and for every 6 months thereafter that the participant is in the study, according to the following scales:
  • Modified Caregiver Strain Index (MCSI)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Morrell, MD, Principal Investigator — NeuroPace, Inc.
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The following data types will be uploaded to the Data Archive for the BRAIN Initiative (DABI):
  * Medical imaging: MRI, CT
  * Neurophysiological recordings: intracranial EEG recordings
  * Data collected from RNS Neurostimulator, reformatted for analysis.
  * Clinical Trial Outcome and Endpoint data.
  * Treatment condition status for subjects.
  Data will be uploaded every 6 months. Access is restricted and must be requested.
Supporting Information: Study Protocol
Time Frame: The dataset and any supporting documentation (including but not limited to the study protocol, statistical analysis plan, and data dictionary) required for the analysis of the data will be made available within one year of the primary publication or within 18 months of the last study visit of the last subject, whichever occurs first.
Access Criteria: Requestors will provide a CV, a description of their resources & facilities, along with a description of their planned analyses. Requests will be evaluated by a Research Review Committee at NeuroPace in accordance with NeuroPace data sharing policies. Approved requests will require execution of a data access agreement based on NeuroPace's existing template.
URL: https://dabi.loni.usc.edu/dsi/UH3NS109557